CLINICAL TRIAL: NCT05319184
Title: Acute Effect of Myofascial Release and Kinesiology Taping on Parameters Associated With Chronic Low Back Pain
Brief Title: Acute Effect of Myofascial Release and Kinesiology Taping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Kubra Kardes, MSc PT, Lecturer, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 003
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Low Back Pain; Kinesio Taping; Myofascial Release Technique
Keywords: Low Back Pain; Kinesio Taping; Myofascial release technique
MeSH Terms: conditions — Low Back Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Myofascial Release Group (Experimental): The application will be made with the patient in the prone position. By applying a few grams of constant force to the lumbar paravertebral muscles bilaterally with the hand of the physiotherapist in the direction of restriction for 3-5 minutes, the fascia will be stretched and allow the tissue to relax on its own. Thus, it is aimed to decrease the tone and stiffness of the paravertebral muscles.
  Interventions: Other: Myofascial Release Technique and Kinesiology Taping
- Kinesiology Taping Group (Experimental): During the application, the participants will be positioned standing and facing backwards due to the ease of application. While taping the lumbar region, the kinesiology tape cut as a long strip (I tape) will be applied paravertebrally to the right and left sides of the spine. Rounded corners will be created to prevent premature loosening and unwanted bends in the belt. The patient will be asked to perform maximum trunk flexion and 2 I-shaped pieces will be taped with 10-15% tension from the lumbar region to the thoracic region. The tape will remain on the patient's skin for 30 minutes.
  Interventions: Other: Myofascial Release Technique and Kinesiology Taping
- Control Group (No Intervention): No intervention.

INTERVENTIONS:
Other: Myofascial Release Technique and Kinesiology Taping — Myofascial release is a manual release technique that increases the elasticity and glide between soft tissue layers, reduces this increased muscle activity and pain intensity. Myofascial release is usually characterized by prolonged mechanical forces exerted directly or indirectly on the limited fascial layers with low load. Following the direction of the fascial restraint, the therapist's hands slowly maintain the stretch and allow the fascia to relax on its own.
  Kinesio Taping is a non-invasive, painless and less time consuming method with fewer side effects. It is an elastic-cotton adhesive tape that is latex-free and can be used on any joint or muscle. It can stretch significantly (130-140% of its original length), which reduces mechanical movement limitations and mimics skin in thickness and elasticity. It is used in the treatment of LBP to reduce muscle tone and stiffness as a rehabilitative taping technique designed to support the body's natural healing process.
  Arms: Kinesiology Taping Group; Myofascial Release Group

SUMMARY:
Chronic low back pain (LBP) is one of the leading causes of activity limitation and disability. The prevalence of chronic CBA among young adults is known to increase, and a recent epidemiological study reported a rate of 42.4% per year among young adults. Studies show that changes in the paravertebral muscles have an important relationship with the formation of Chronic LBP, and therefore, evaluation of the mechanical properties of the paravertebral muscles is of great importance for the clinical diagnosis and treatment of Chronic LBP.

Mechanical properties of the muscle, such as muscle stiffness and tone, are considered essential for maintaining efficient muscle contraction. Abnormally high muscle tone blocks blood flow, leading to faster muscle fatigue and slower muscle recovery. When there is abnormally high muscle stiffness, stretching the stiffened antagonist muscles requires more effort, resulting in lower exercise efficiency. Muscle stiffness is one of the critical indicators of energy storage of the muscle-tendon unit, which has a significant effect on the control of joint movement. Altered tone and stiffness in the lumbar myofascial region have been described in association with underlying pathologies and symptoms in people with Chronic LBP. Rehabilitation interventions such as manual therapy or therapeutic exercises are common techniques for the treatment of chronic Chronic LBP because of their benefits in altering muscle tone and stiffness by reducing paraspinal muscle activity.

Although the effectiveness of the myofascial release technique in individuals with Chronic LBP is supported in the literature, the long-term use of the therapist's hand support creates difficulties in practice in the clinical setting. The KT technique, on the other hand, seems to be a method that can be used as an alternative to myofascial release technique in the treatment of Chronic LBP, since it is an easy-to-use and time-consuming approach. When the studies conducted to date are examined, no study has been found that compares the effectiveness of myofascial release and kinesiology taping applied to individuals with Chronic LBP. The aim of our study is to compare the acute effect of myofascial release and kinesiology taping in individuals with Chronic LBP.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-45
* Being diagnosed with nonspecific chronic low back pain (lasting longer than 3 months)
* Volunteering to participate in the study

Exclusion Criteria:

* Those who have had major surgery or trauma related to the musculoskeletal system, especially the lumbar region
* Those with neurological disease
* Those with rheumatic disease in the active period
* Those with systemic diseases (Diabetes, hypothyroidism, infection, malignancy...)
* Those with serious psychological problems (BDI score of 30 and above)
* Those with kinesiology tape allergies
* Those with contraindications to myofascial release therapy (acute inflammations, viral and bacterial infections, infectious diseases, fever, deep vein thrombosis, active malignant disease, aneurysms)
* Those who received physiotherapeutic intervention to the lumbar region in the last 6 months
* Obesity (BMI≥30 kg/m2)
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Muscle Tone and Stiffness | 4 weeks
  Muscle tone and stiffness will be evaluated with a myotonometer. The myotonusometer was developed for the objective measurement of mechanical muscle properties. Myotonusometry reflects the viscoelastic properties of the muscle such as tone and stiffness by creating oscillation in the muscle fiber and is an acceptable and reliable method for measuring the mechanical properties of the muscle in young adults with chronic LBP. The device measures muscle tone as the natural oscillation frequency (Hz) calculated as Hz = 1/T; where T is the oscillation time measured in seconds. Muscle stiffness (N/m) is related to the maximum acceleration of oscillation and tissue deformation recorded by the transducer.
Visual Analogue Scale | 4 weeks
  The Visual Analog Scale is a simple, precise and reproducible tool that is often used to assess pain severity. Due to its easy application, it is one of the most frequently used measurement tools to measure the severity of pain in low back pain. It consists of a horizontal or vertical line ten cm long. The starting point of the line, '0', represents no pain, and the ending point, '10', represents the most severe pain imaginable. Pain intensity increases as you go from 0 to 10. The patient is asked to mark the severity of the pain on the line, the point marked by the patient is recorded in cm.
Joint Range of Motion | 4 weeks
  Lumbar region flexion, extension, lateral flexion and rotation movements will be measured bilaterally with a digital goniometer. Measurements will be repeated 3 times and the average value will be recorded in degrees.

SECONDARY OUTCOMES:
Mobility | 4 weeks
  The Modified Schober Test will be used to evaluate the mobility of the lumbar region. For this test, while the patient is standing, mark 10 cm upwards from the second sacral spinous process and 5 cm downwards from this protrusion (the distance between the two points is 15 cm). The patient has maximum flexion of the trunk and the distance between the two points is measured. The difference is found by subtracting 15 cm (the distance between two points in upright posture) from the value found. The fact that this difference is less than 5 cm indicates that the mobility of the lumbar region is reduced.
Progressive İsoinartial Lifting Evaluation | 4 weeks
  The PILE Test will be used to evaluate the general body strength and endurance of the participants. Application of the test: The test starts with a weight of 3.6 kg for women and 5.9 kg for men. These weights are put into the box and the participants are asked to lift this box to a 75 cm high table 4 times within 20 seconds. After each completed lap, a weight of 2.25 kg for women and 4.5 kg for men is added to the box. If the participant fails to complete 4 repetitions within 20 seconds, wishes to discontinue the test due to fatigue or extreme discomfort (psychophysical endpoint), reaches 85% of maximum heart rate (220-years), or reaches the maximum weight that can be safely lifted (55-60% of body weight) i) the test is terminated. The maximum weight lifted and the number of repetitions are recorded. By multiplying the maximum weight lifted and the number of repetitions, the total work done is calculated and recorded.
1 Minute Stepping Test | 4 weeks
  The step test will be used to evaluate the physical performance of the participants. During the test, participants will be asked to go up and down a step of 40 cm for 1 minute. The number of repetitions performed in 1 minute will be recorded for the right and left sides.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul university Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No